CLINICAL TRIAL: NCT00793286
Title: Stapler Versus Glue for Laparoscopic Groin Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Guido Beldi, MD, Dep. of Visceral and Transplantsurgery, Bern University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEK_89_04
Record Dates: First submitted 2008-11-18; First posted 2008-11-19 (Estimated); Last update posted 2008-11-24 (Estimated); Status verified 2008-11

CONDITIONS: Inguinal Hernia; Recurrence; Pain
Keywords: inguinal hernia; laparoscopy; mesh
MeSH Terms: conditions — Hernia, Inguinal; Recurrence; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): Mesh fixation by staples
  Interventions: Procedure: Mesh fixation by staples
- B (Other): Mesh fixation by glue
  Interventions: Procedure: Mesh fixation by glue

INTERVENTIONS:
Procedure: Mesh fixation by staples — Mesh fixation by staples
  Arms: A
Procedure: Mesh fixation by glue — Mesh fixation by glue
  Other Names: N-Butyl-2 Cyanoacrulat Glue
  Arms: B

SUMMARY:
Repair of inguinal hernia is the most common operation of the general surgeon. In recent years, it was recognized that chronic postoperative pain is as important for postoperative outcome as recurrent hernia. The incidence of pain or discomfort ranges up to 60% of operated patients. Despite the fact that laparoscopic hernia repair has been shown to reduce postoperative pain compared to open hernia repair, up to 5% of patients suffer from persistent discomfort. During that operation the mesh is either fixed using a stapler or tissue adhesive glue. With the current study we compare postoperative pain between patients undergoing laparoscopic inguinal hernia repair with either mesh fixation using a stapler or tissue adhesive. The use of von Frey monofilaments allows to describe pain with a high sensitivity.

DETAILED DESCRIPTION:
Despite the fact that laparoscopic hernia repair has been shown to reduce postoperative pain compared to open hernia repair, up to 5% of patients suffer from persistent discomfort. During that operation the mesh is either fixed using a stapler or tissue adhesive glue. With the current study we compare postoperative pain between patients undergoing laparoscopic inguinal hernia repair with either mesh fixation using a stapler or tissue adhesive. The use of von Frey monofilaments allows to describe pain with a high sensitivity.

To perform a prospective randomized trial comparing pain after inguinal hernia repair using either fixation with stapler or histoacryl.

The standard TAPP procedure is performed under general anesthesia. Patients receive a single shot antibiotic prophylaxis, using Amoxicillin/Clavulanic Acids. Operations are performed by resident surgeons under supervision, consultants or senior consultants. After hernial sac dissection and retraction, preperitoneal fat is removed bluntly and Cooper's ligament is identified. A Vypro II ® (Ethicon ®) prosthetic mesh, 10x15 cm, is placed and fixed depending on randomization with either 5 mm Protack TM (Autosuture TM) or Glubran ® 2 (G.E.M., Viareggio, Italy). Randomization is performed in permutated block of 20 using sealed envelopes. Where tissue glue is used, meshs are additionally fixed caudally and laterocaudally. Peritoneal closure over the mesh is performed using resorptive sutures. Glubran ® 2 is a cyanoacrylate tissue adhesive. Follow up assessment: The use of analgesics in the postoperative period is standardized using paracetamol and morphine derivates. Following discharge patients are liberated of physical restrictions. Patient follow-up will be performed after 6 weeks, 6 and 12 months postoperatively. Patients are advised to mention pain in the operated groin area. In addition the Visual Analogue Scale is used to evaluate pain intensity.Statistical comparison is done using Mann-Whitney Test and Chi square Test (significance p < 0,05).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for laparoscopic primary inguinal hernia repair
* uni- or bilateral patients with recurrent hernias after anterior surgical technique
* written informed consent

Exclusion Criteria:

* general contradictions for laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2004-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Recurrence | 6 weeks, 6 months, 12 months postoperative

SECONDARY OUTCOMES:
postoperative pain | 6 weeks, 6 months, 12 months postoperative
sensibility disorder | 6 weeks, 6 months, 12 months postoperative
intra- and postoperative complications | 6 weeks, 6 months, 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Guido Beldi, MD, Principal Investigator — Dep. of Visceral and Transplantsurgery, Bern University Hospital
Locations (1):
- Dep. of Visceral and Transplantsurgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] McCormack K, Scott NW, Go PM, Ross S, Grant AM; EU Hernia Trialists Collaboration. Laparoscopic techniques versus open techniques for inguinal hernia repair. Cochrane Database Syst Rev. 2003;2003(1):CD001785. doi: 10.1002/14651858.CD001785. PMID 12535413
- [Background] Cunningham J, Temple WJ, Mitchell P, Nixon JA, Preshaw RM, Hagen NA. Cooperative hernia study. Pain in the postrepair patient. Ann Surg. 1996 Nov;224(5):598-602. doi: 10.1097/00000658-199611000-00003. PMID 8916874
- [Background] Bay-Nielsen M, Perkins FM, Kehlet H; Danish Hernia Database. Pain and functional impairment 1 year after inguinal herniorrhaphy: a nationwide questionnaire study. Ann Surg. 2001 Jan;233(1):1-7. doi: 10.1097/00000658-200101000-00001. PMID 11141218
- [Background] Laparoscopic versus open repair of groin hernia: a randomised comparison. The MRC Laparoscopic Groin Hernia Trial Group. Lancet. 1999 Jul 17;354(9174):185-90. PMID 10421299
- [Background] Katkhouda N, Mavor E, Friedlander MH, Mason RJ, Kiyabu M, Grant SW, Achanta K, Kirkman EL, Narayanan K, Essani R. Use of fibrin sealant for prosthetic mesh fixation in laparoscopic extraperitoneal inguinal hernia repair. Ann Surg. 2001 Jan;233(1):18-25. doi: 10.1097/00000658-200101000-00004. PMID 11141220
- [Background] Jourdan IC, Bailey ME. Initial experience with the use of N-butyl 2-cyanoacrylate glue for the fixation of polypropylene mesh in laparoscopic hernia repair. Surg Laparosc Endosc. 1998 Aug;8(4):291-3. PMID 9703604
- [Background] Neumayer L, Giobbie-Hurder A, Jonasson O, Fitzgibbons R Jr, Dunlop D, Gibbs J, Reda D, Henderson W; Veterans Affairs Cooperative Studies Program 456 Investigators. Open mesh versus laparoscopic mesh repair of inguinal hernia. N Engl J Med. 2004 Apr 29;350(18):1819-27. doi: 10.1056/NEJMoa040093. Epub 2004 Apr 25. PMID 15107485
- [Background] Bittner R, Schmedt CG, Schwarz J, Kraft K, Leibl BJ. Laparoscopic transperitoneal procedure for routine repair of groin hernia. Br J Surg. 2002 Aug;89(8):1062-6. doi: 10.1046/j.1365-2168.2002.02178.x. PMID 12153636